CLINICAL TRIAL: NCT01993147
Title: Functional Differences in Effortful Control
Acronym: FDEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Behavioral manipulation failed so the trial did not occur
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chandra Sekhar Sripada, Chandra Sekhar Sripada, MD, PhD, Dept. of Psychiatry, UofM, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-MED-HUM00074465
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Methylphenidate; Placebo; functional Magnetic Resonance Imaging (fMRI); Attention Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual Task Paradigm (Other): This arm does not involve any drug intervention, it is an experimental type consisting of 80 subjects to study the dual task paradigm implemented during the fMRI scanning session. 80 subjects will perform the fMRI scan but will not undergo any drug intervention.
  Interventions: Behavioral: Dual task paradigm pilot

INTERVENTIONS:
Behavioral: Dual task paradigm pilot

SUMMARY:
The purpose of this study was to learn more about the brain circuits involved with effortful control in healthy adult participants. It was planned that the study would enroll 80 participants to a dual task paradigm pilot while undergoing a fMRI scan to assess brain mechanisms that cause the "depletion effect". This effect refers to the observation that people perform more poorly on effortful control tasks after they have already performed task requiring effortful control. Then subsequent study participants would be given either methylphenidate (also known as 'Ritalin') which is FDA approved and the most widely-used medication for Attention Deficit Hyperactivity Disorder (ADHD) or a placebo, which is a sugar pill. Each participant would also perform some computer tasks that have been shown in previous studies to require effortful control while undergoing an fMRI (functional Magnetic Resonance Imaging) which takes a special kind of picture of the brain. The study's goal was to learn more about the brain mechanisms by which methylphenidate improves effortful control. After enrolling the first 50 participants, the study assessed whether a depletion effect was observed in the dual task paradigm. It was found that there was not: there was no statistically significant difference in effortful control performance comparing subjects who did and did not perform a prior effortful control task. Because the behavioral manipulation failed, it was determined that the drug manipulation portion of the study was no longer justified. Thus, after enrolling 50 participants to the pilot part of the study, the decision was made to terminate the study without beginning the trial of methylphenidate.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness

Exclusion Criteria:

* Any clinically significant personal or family history of cardiac problems
* Any current Axis I psychiatric disorder (diagnosis as verified by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-IV)
* A previous adequate trial with methylphenidate (Ritalin)
* Currently taking any psychoactive medications
* Any clinically significant medical condition
* Any clinically significant neurological problem (seizures, tics, serious head injury)
* Contraindications to MRI (metal objects in body or claustrophobia)
* Currently pregnant or lactating
* Alcohol or substance abuse (current or in the past 2 years)
* Left-handedness or ambidextrous
* Liver or kidney disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2015-06-08 (Actual); Study Completion 2015-06-08 (Actual)

PRIMARY OUTCOMES:
Reaction Time on the Multi-Source Interference Task | 3 hours

SECONDARY OUTCOMES:
Accuracy on the Multi-Source Interference Task | 3 hours
  Accuracy is the calculated percentage of correct responses over total trials
Reaction time variability on the Multi-Source Interference Task | 3 hours
  Reaction Time Variability is the standard deviation of the trial to trial reaction time distribution (the standard deviation is a unitless quantity) on the Multi-Source Interference Task.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Sekhar Sripada, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- Rachel Upjohn Building, East Medical Campus, Ann Arbor, Michigan, United States